CLINICAL TRIAL: NCT03697902
Title: Influence of Imaging Angle in Measurement of Cisterna Magna in the Second Trimester
Brief Title: Influence of Imaging Angle in Measurement of Cisterna Magna
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med Flavio Hernández Castro, Principal investigator MD PhD Flavio Hernández Castro, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GI19-00010
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-10

CONDITIONS: Fetal Cisterna Magna Length; Ultrasonography
Keywords: Cisterna magna length; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonographic Measurement on Fetal cisterna magna length — The length measurement on the fetal cisterna magna (CM) with an angle of 0° between the transducer and the axial cerebellar plane of the fetal head (midline structures will be perpendicular to the ultrasound beam). After that, CM will be measured again after moving the transducer approximately 30° towards the fetal occiput.
  Measurements will be performed on the axial cerebellar plane using internal landmarks including the cavum septi pellucidi, thalamus, third ventricle, cerebral peduncles and cerebellar hemispheres.The anteroposterior measurement will be made between the posterior border of the cerebellar vermis and the internal face of the occipital bone.
  All the ultrasonography examinations were performed abdominally, using 3-5 megahertz (MHz) transducers.

SUMMARY:
The aim of this study is to determine the effect of imaging angle on the measurement of fetal cisterna magna (CM) in the second trimester.

Fetal CM will be prospectively measured in women at 18-24.6 weeks' gestation. Measurements will be made on different angles between the transducer and fetal cerebellar axial plane with internal landmarks.

Design: Observative, cross sectional

DETAILED DESCRIPTION:
Patients and methods: women with low risk single pregnancy will be studied. Fetuses with multiple pregnancies, maternal chronic disease and severe congenital anomalies except mega cisterna magna (MCM) will be excluded from the study. Measurements will be performed on the axial cerebellar plane.The anteroposterior measurement will be made between the posterior border of the cerebellar vermis and the internal face of the occipital bone.

The primary outcome variables will be cisterna magna length measured on different angles between the transducer and the axial cerebellar plane of the fetal head.

Cisterna magna length measurement related to fetal presentation and gender will be secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the 18th and 24th weeks.
* Confirmed gestational age by regular menstrual cycle or determined from crown- rump length at first trimester ultrasonography for those with unknown menstruation date .

Exclusion Criteria:

* Uncertain gestational age
* Twin or multiple pregnancy.
* Increased risk for aneuploidy determined by first trimester screening.
* Absence of intracranial translucency in first trimester ultrasound examination.
* Fetal malformations identified EXCEPT megacisterna magna.
* Karyotype anomaly.
* Chronic maternal diseases such as arterial hypertension, diabetes mellitus, hypothyroidism and hyperthyroidism.
* Failure to obtain accurate measurement for technical reasons.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with low risk pregnancy between the 18th and 24th weeks with confirm gestational age who wil be referred to our prenatal diagnosis unit for ultrasonography to be performed in their second trimester.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Cisterna Magna length | 24 hours
  The length measurement on the CM with an angle of 0° between the transducer and the axial cerebellar plane of the fetal head (midline structures will be perpendicular to the ultrasound beam). After that, CM will be measured again after moving the transducer approximately 30° towards the fetal occiput. Measurements of the anteroposterior diameter Will be obtained along straight lines between the posterior border of the cerebellar vermis and the internal face of the occipital bone.

SECONDARY OUTCOMES:
Cisterna Magna length according to fetal presentation | 24 hours
  The length measurement on the CM with an angle of 0° between the transducer and the axial cerebellar plane of the fetal head (midline structures will be perpendicular to the ultrasound beam). After that, CM will be measured again after moving the transducer approximately 30° towards the fetal occiput. Measurements will be made in fetuses with cephalic and breech presentation. Another measurement will be made in fetuses with cephalic presentation that had converted to breech presentation or viceversa in less than 24 hours.
Cisterna Magna length according to fetal sex | 24 hours
  The length measurement on the cisterna magna (CM) with an angle of 0° between the transducer and the axial cerebellar plane of the fetal head (midline structures will be perpendicular to the ultrasound beam). After that, CM will be measured again after moving the transducer approximately 30° towards the fetal occiput. Those measurements will be compare between male and female fetuses.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Hernández-Castro, Dr. med, Principal Investigator — Hospital Universitario Dr. José Eleuterio González UANL
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho JY, Kim KW, Lee YH, Toi A. Measurement of nuchal skin fold thickness in the second trimester: influence of imaging angle and fetal presentation. Ultrasound Obstet Gynecol. 2005 Mar;25(3):253-7. doi: 10.1002/uog.1847. PMID 15736211
- [Background] Araujo Junior E, Martins WP, Rolo LC, Pires CR, Zanforlin Filho SM. Normative data for fetal cisterna magna length measurement between 18 and 24 weeks of pregnancy. Childs Nerv Syst. 2014 Jan;30(1):9-12. doi: 10.1007/s00381-013-2298-y. PMID 24122018
- [Background] Serhatlioglu S, Kocakoc E, Kiris A, Sapmaz E, Boztosun Y, Bozgeyik Z. Sonographic measurement of the fetal cerebellum, cisterna magna, and cavum septum pellucidum in normal fetuses in the second and third trimesters of pregnancy. J Clin Ultrasound. 2003 May;31(4):194-200. doi: 10.1002/jcu.10163. PMID 12692827
- [Background] Liu Z, Han J, Fu F, Liu J, Li R, Yang X, Pan M, Zhen L, Li D, Liao C. Outcome of isolated enlarged cisterna magna identified in utero: experience at a single medical center in mainland China. Prenat Diagn. 2017 Jun;37(6):575-582. doi: 10.1002/pd.5046. Epub 2017 May 10. PMID 28370151